CLINICAL TRIAL: NCT00152061
Title: The Role of 3TC/FTC in Partially Suppressive Antiretroviral Regimens: The Switch Study
Brief Title: The Switch Study: The Role of Lamivudine/Emtricitabine (3TC/FTC) in Antiretroviral Regimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Health & Hospital System (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 74009; IRB protocol 74009; SPO number 25036
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: HIV Infections
Keywords: HIV; Antiretroviral Drug Resistance; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Racivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 3TC and FTC

SUMMARY:
In this study the researchers will be enrolling patients who are failing their current antiretroviral regimen who also have resistance to 3TC or FTC. Patients will have their current antiretroviral regimen changed based on resistance testing and also be randomly assigned to either include, or not include 3TC/FTC in this new regimen. The purpose of the research is to investigate whether the change in therapy results in a decrease in the amount of virus particles and an increase in the CD4 cell count. In addition the researchers are investigating the relationship between the existence of resistance and the rate of decrease in viral load, and also to determine if continuing 3TC/FTC (despite being resistant to the medications) has any effect on the rate of decrease of viral load, or effect on CD4 counts.

DETAILED DESCRIPTION:
In this randomized, open-label, controlled trial, HIV-infected patients who are failing 3TC/FTC-containing highly active antiretroviral therapy, (HAART), will be offered individual treatment selection based on best clinical judgment and genotypic HIV-RNA resistance analysis. Patients who meet entry criteria will first be randomized to either continue or discontinue 3TC/FTC while they remain on their current therapy. HIV-1 viral load will be measured 4 times over a period of 14 days to determine the virologic response to this change. At day 14, each patient's regimen will be optimized to a new combination based on a genotype test taken at study entry. Patients will then start on the new salvage regimen, including or not including 3TC/FTC based on their initial randomization. Additional HIV-1 viral load measurements will be obtained to determine the virologic response to the new salvage regimen over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive patients >= 18 years of age
* Willingness and ability to understand and sign a written informed consent and comply with the protocol procedure
* Prior treatment with nucleoside reverse transcriptase inhibitors (NRTI's), non-nucleoside reverse transcriptase inhibitors (NNRTI's) and protease inhibitor (PI)-containing regimens
* On a stable PI and 3TC or FTC -containing regimen for >= 2 months
* Plasma HIV-1 RNA >5000 copies/ml
* CD4 >100
* Documented M184V or I on genotype within 3 months of study entry
* At least 3 PI-associated resistance mutations on genotype within 3 months of study entry, (including known resistance mutations at codons 10, 30, 46, 50, 54, 71, 82, 84, and 90)

Exclusion Criteria:

* In the opinion of the investigator a patient that is either unwilling or unable to be adherent to antiretroviral drugs
* Requirement for concomitant treatment with medicines that interfere with the therapy prescribed in the study
* Patients who have never taken 3TC or FTC, or with no prior documentation of the M184V mutation
* Active hepatitis B infection
* Vaccination within 2 weeks of entering the study
* An acute opportunistic illness within 4 weeks of entering the study; chronic infections will not be excluded
* Use of immunomodulatory medications such as IL-2
* Planned use of enfuvirtide, (T20) in salvage regimen, (in T20 naïve subjects)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-01; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the role of lamivudine, (3TC), and emtricitabine, (FTC), in salvage regimens in patients with prior 3TC/FTC use, documented resistance to 3TC/FTC, and ongoing viremia as assessed by:
Impact on the initial rate of change in HIV-1 viral load after removing 3TC/FTC from the failing regimen, and
Overall change from baseline in HIV-1 viral load at 24 weeks (HIV-VL AUC 24 wks).

SECONDARY OUTCOMES:
To evaluate the impact of continued versus discontinued 3TC/FTC on the prevalence, frequency and dynamics of the M184V/I amino acid substitution over 24 weeks.
To determine the proportion of patients failing and/or not responding to therapy after 24 weeks as defined by failure to achieve HIV-1 viral load less than 400 copies/ml and/or less than 50 copies/ml
To assess the changes from baseline in absolute CD4 (and CD8) cell counts at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zolopa, MD, Principal Investigator — Stanford University
Locations (1):
- Santa Clara Medical Center, PACE Clinic, San Jose, California, United States